CLINICAL TRIAL: NCT04259554
Title: Orbitofrontal Cortex Transcranial Magnetic Stimulation in Patients With Emotionally Unstable Personality Disorder and Depression
Brief Title: OFC rTMS in Emotionally Unstable and Depressed Patients
Acronym: ORIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1615-101
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Personality Disorder, Borderline; Personality Disorder; Unstable; Depression
Keywords: rTMS
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OFC rTMS (Experimental): repetitive transcranial magnetic stimulation
  Interventions: Device: OFC rTMS

INTERVENTIONS:
Device: OFC rTMS — repetitive transcranial magnetic stimulation over right orbito-frontal cortex with 1Hz (360 pulses in 6 trains á 60 pulses with 30s intertrain-interval)

SUMMARY:
Treatment of depression with conventional transcranial magnetic stimulation (rTMS) has shown high evidence using high-frequency left dorsolateral prefrontal cortex (DLPFC) stimulation. Recently, it could be demonstrated that treatment of the right orbitofrontal cortex may be effective in patients who did not respond to conventional DLPFC rTMS. Orbitofrontal cortex (OFC) seem to be involved in the etiopathology of emotionally instable personality disorders. Thus, the present one-arm trial is a pilot study investigating if OFC rTMS is feasable, tolerable and effective.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10: F60.30 or F60.31
* depressive symptoms and HAMD-21 score of at least 7
* sex: female and male
* residence in Germany and German speaking
* written informed consent

Exclusion Criteria:

* meeting the contraindications for transcranial magnetic stimulation (electric devices or metal implants in the body, e.g. cardiac pace maker, insulin pump)
* neurological disorders (e.g. cerebrovascular events, neurodegenerative disorder, epilepsy, brain malformation, severe head trauma)
* participation in another study parallel to the Trial
* other mental or somatic illness which is not compatible with participation according to the principal investigator
* pregnancy or breastfeeding period
* psychiatric confinement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Hamilton depression rating scale (HDRS) | 4 weeks
  measurment of depressivity: 21 items with a range 0-65 and higher values indicating higher scores

SECONDARY OUTCOMES:
Major Depression Inventory (MDI) | 2 weeks, 4 weeks, 12 weeks
  measurment of depressivity: 10 items with a range 0-50 and higher values indicating higher scores
Clinical global impression (CGI) | 2 weeks, 4 weeks, 12 weeks
  measure of overall symptom severity and treatment response on a scale 1-7 with higher scores presenting more symptoms
Depression module of the Patient health questionnaire (PHQ-D) | 4 weeks, 12 weeks
  measurment of depressivity: 9 items with a range 0-27 and higher values indicating higher scores
Barratt impulsiveness Scale (BIS) | 4 weeks, 12 weeks
  measurment of impulsivity: 30 items with a range 0-120 and higher values indicating higher scores
Numeric rating scale of pain | 2 weeks, 4 weeks
  Numeric rating scale of pain (the higher the score the higher the pain) with a range 0-10
nicotine use | 2 weeks, 4 weeks, 12 weeks
  number of smoked cigarettes per day (the higher the value the higher the use)
Hamilton depression rating scale (HDRS) | 2 weeks, 4 weeks, 12 weeks
  measurment of depressivity: 21 items with a range 0-65 and higher values indicating higher scores
Borderline Symptom List (BSL-23) | 2 weeks, 4 weeks, 12 weeks
  measurment of symptoms of borderline personality disorder: 23 items with a range 0-92 and higher values indicating higher scores

CONTACTS AND LOCATIONS:
Locations (1):
- University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No